CLINICAL TRIAL: NCT04008420
Title: The Association of Intraoperative Oxygen Reserve Index and Postoperative Pulmonary Complications in Robot-assisted Esophagectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2019-0448
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Endotracheal Intubation; Robotic Esophagectomy; Esophagectomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults who are scheduled to undergo robotic esophagectomy: Adults who are scheduled to undergo robotic esophagectomy
  Interventions: Other: monitoring of the oxygen reserve index

INTERVENTIONS:
Other: monitoring of the oxygen reserve index — The investigators will enroll adult patients who will undergo robotic esophagectomy under general anesthesia. The oxygen reserve index will be monitored continuously during anesthesia. The postoperative complications will be recorded after surgery.

SUMMARY:
The World Health Organization (WHO) has proposed the use of 80% high-dose inhalation oxygen (FiO2) during surgery to reduce postoperative infection in adult patients undergoing general anesthesia. However, high-dose inhaled oxygen increases the risk of oxygen toxicity by increasing reactive oxygen species, and according to a recent research, hyperoxia in the ICU is one of the causes of mortality. In patients with general anesthesia requiring intubation, high-dose inhaled oxygen was associated with postoperative pulmonary complications in a dose-proportional manner and was significantly associated with mortality within 30 days after surgery. Therefore, it is necessary to study the optimum oxygen concentration during surgery to reduce postoperative pulmonary complications in general anesthesia patients who require intubation. Esophagectomy for esophageal cancer still has higher morbidity and mortality rates than other common procedures. There are several factors such as aneurysmal leakage, esophageal substitute necrosis, cardiac complications, and pulmonary complications. Pulmonary complications have been reported to be a very important factor. Therefore, various methods have been proposed to reduce pulmonary complications after esophageal cancer surgery. One of them is minimally invasive surgery. However, even in the case of a thoracoscopic operation using a robot, one lung ventilation is inevitable for securing the visual field during surgery, and hypoxia and hyperoxia are known to be associated with postoperative acute lung injury. Therefore, in order to reduce postoperative pulmonary complications in the esophagectomy using robots, it is necessary to study the optimum oxygen concentration during surgery. The recently developed oxygen reserve index (ORI) uses a non-invasive sensor attached to the finger, similar to pulse oximetry, to detect persistent hyperoxia of more than 100 mmHg and less than 200 mmHg. Therefore, if the oxygen reserve index is used for robotic esophagectomy, which requires one lung ventilation, the degree of oxygenation of the patient can be monitored continuously and accurately. The authors will measure the oxygen reserve index in robotic esophagectomy, and analyze the correlation between oxygen reserve index and postoperative pulmonary complications. Furthermore, the cut-off value of the oxygen reserve index, which can reduce pulmonary complications, will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adults who are scheduled to undergo robotic esophagectomy

Exclusion Criteria:

* 1. Patients under 20 years old
* 2. Patients who can not read the consent form or are not fluent in Korean
* 3. Patients who refused the clinical trial
* 4. Patients admitted to the intensive care unit with endotracheal tube

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who are scheduled to undergo robotic esophagectomy
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-07-31 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
The value of oxygen reserve index during anesthesia | Participants will followed until discharge (within about 2 months after surgery).
  The investigators will monitor the oxygen reserve index during anesthesia.

SECONDARY OUTCOMES:
Postoperative pulmonary complications | Participants will followed until discharge (within about 2 months after surgery).
  The investigators will observe and record the occurrence of the postoperative pulmonary complications.

CONTACTS AND LOCATIONS:
Overall Officials: So Yeon Kim, MD, Principal Investigator — Severance Hospital
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institue, Yonsei Universiy College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No